CLINICAL TRIAL: NCT02906930
Title: Efficacy and Safety of Oral Semaglutide Versus Placebo in Subjects With Type 2 Diabetes Mellitus Treated With Diet and Exercise Only.
Acronym: PIONEER 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4233; 2015-005622-19 (EudraCT Number); U1111-1177-5112 (Other: WHO); JapicCTI-163384 (Other: JapicCTI)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 3 mg oral semaglutide (Experimental)
  Interventions: Drug: semaglutide
- 7 mg oral semaglutide (Experimental)
  Interventions: Drug: semaglutide
- 14 mg oral semaglutide (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Oral administration once daily.
  Arms: 14 mg oral semaglutide; 3 mg oral semaglutide; 7 mg oral semaglutide
Drug: placebo — Oral administration once daily.
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate efficacy and safety of oral semaglutide versus placebo in subjects with type 2 diabetes mellitus treated with diet and exercise only.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - Male or female, age above or equal to 18 years at the time of signing informed consent.For Japan only: Male or female, age above or equal to 20 years at the time of signing informed consent. For Algeria only: Male or female, age above or equal to 19 years at the time of signing informed consent - Diagnosed with type 2 diabetes mellitus for at least 30 days prior to day of screening - HbA1c (glycosylated haemoglobin) between 7.0-9.5% (53-80 mmol/mol) (both inclusive) - Treatment with diet and exercise for at least 30 days prior to day of screening Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice) For Japan only: Adequate contraceptive measures are abstinence (not having sex), diaphragm, condom (by the partner), intrauterine device, sponge, spermicide or oral contraceptives.For Czech Republic only: Adequate contraceptive measures are always one highly reliable method (such as intrauterine device, sterilisation of one of the partners, hormonal birth control methods) plus one supplementary barrier method (such as condom, diaphragm) with a spermicide. In justified cases, this combination may be replaced with a double-barrier method with a spermicide. Total sexual abstinence may also be considered contraception. (Please note: hormonal contraception should always be discussed with a gynaecologist) - Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol - Family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinomas - History of pancreatitis (acute or chronic) - History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) - Any of the following: myocardial infarction, stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation - Subjects presently classified as being in New York Heart Association Class IV. - Planned coronary, carotid or peripheral artery revascularisation known on the day of screening - Subjects with alanine aminotransferase above 2.5 x upper normal limit - Renal impairment defined as estimated glomerular filtration rate below 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula - Treatment with any medication for the indication of diabetes or obesity in a period of 90 days before the day of screening. An exception is short-term insulin treatment for acute illness for a total of below or equal to 14 days - Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation - History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in-situ carcinomas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (82):
- United States (51):
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, North Hollywood, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Jose, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Doral, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Spring Hill, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Woodstock, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Nampa, Idaho
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Rochester, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Elkhorn, Nebraska
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Willoughby Hills, Ohio
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, Bountiful, Utah
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Salem, Virginia
- Novo Nordisk Investigational Site, Algiers, Algeria
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Czechia (5):
  - Novo Nordisk Investigational Site, Broumov
  - Novo Nordisk Investigational Site, Chrudim
  - Novo Nordisk Investigational Site, Mladá Boleslav
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Prague
- Italy (5):
  - Novo Nordisk Investigational Site, Como
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Pisa
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Siena
- Japan (3):
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yokohama-shi, Kanagawa
- Mexico (2):
  - Novo Nordisk Investigational Site, Ciudad Madero, Tamaulipas
  - Novo Nordisk Investigational Site, Aguascalientes
- Romania (3):
  - Novo Nordisk Investigational Site, Târgovişte, Dâmbovița County
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Bucharest
- Russia (8):
  - Novo Nordisk Investigational Site, Dzerzhinskiy
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Yaroslavl
  - Novo Nordisk Investigational Site, Yoshkar-Ola
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Background] Kolotkin RL, Williams VSL, Ervin CM, Williams N, Meincke HH, Qin S, von Huth Smith L, Fehnel SE. Validation of a new measure of quality of life in obesity trials: Impact of Weight on Quality of Life-Lite Clinical Trials Version. Clin Obes. 2019 Jun;9(3):e12310. doi: 10.1111/cob.12310. Epub 2019 Apr 16. PMID 30993900
- [Background] Aroda VR, Saugstrup T, Buse JB, Donsmark M, Zacho J, Davies MJ. Incorporating and interpreting regulatory guidance on estimands in diabetes clinical trials: The PIONEER 1 randomized clinical trial as an example. Diabetes Obes Metab. 2019 Oct;21(10):2203-2210. doi: 10.1111/dom.13804. Epub 2019 Jun 30. PMID 31168921
- [Result] Aroda VR, Rosenstock J, Terauchi Y, Altuntas Y, Lalic NM, Morales Villegas EC, Jeppesen OK, Christiansen E, Hertz CL, Haluzik M; PIONEER 1 Investigators. PIONEER 1: Randomized Clinical Trial of the Efficacy and Safety of Oral Semaglutide Monotherapy in Comparison With Placebo in Patients With Type 2 Diabetes. Diabetes Care. 2019 Sep;42(9):1724-1732. doi: 10.2337/dc19-0749. Epub 2019 Jun 11. PMID 31186300
- [Result] Araki E, Terauchi Y, Watada H, Deenadayalan S, Christiansen E, Horio H, Kadowaki T. Efficacy and safety of oral semaglutide in Japanese patients with type 2 diabetes: A post hoc subgroup analysis of the PIONEER 1, 3, 4 and 8 trials. Diabetes Obes Metab. 2021 Dec;23(12):2785-2794. doi: 10.1111/dom.14536. Epub 2021 Sep 27. PMID 34472698
- [Result] Aroda VR, Bauer R, Christiansen E, Haluzik M, Kallenbach K, Montanya E, Rosenstock J, Meier JJ. Efficacy and safety of oral semaglutide by subgroups of patient characteristics in the PIONEER phase 3 programme. Diabetes Obes Metab. 2022 Jul;24(7):1338-1350. doi: 10.1111/dom.14710. Epub 2022 May 9. PMID 35373893
- [Result] Gorst-Rasmussen A, Tarp-Johansen MJ. Fast tipping point sensitivity analyses in clinical trials with missing continuous outcomes under multiple imputation. J Biopharm Stat. 2022 Nov 2;32(6):942-953. doi: 10.1080/10543406.2022.2058525. Epub 2022 Jun 2. PMID 35653556
- [Derived] Mosenzon O, Capehorn MS, De Remigis A, Rasmussen S, Weimers P, Rosenstock J. Impact of semaglutide on high-sensitivity C-reactive protein: exploratory patient-level analyses of SUSTAIN and PIONEER randomized clinical trials. Cardiovasc Diabetol. 2022 Sep 2;21(1):172. doi: 10.1186/s12933-022-01585-7. PMID 36056351
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 93 sites in 9 countries as follows: Algeria: 4 sites screened/4 sites randomised subjects; Bulgaria: 3/3; Czech Republic: 5 /5; Japan: 6/6; Mexico: 2/2; Russian Federation: 9/9; Serbia: 3/3; Turkey: 7/7; United States: 53/48.
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 3 mg: Participants were to take oral semaglutide 3 mg tablets once daily from week 0 to week 26.
- Oral Semaglutide 7 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 26: 3 mg from week 0 to week 4 and 7 mg from week 4 to week 26.
- Oral Semaglutide 14 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 26: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 26.
- Placebo: Participants were to take placebo tablets once daily for a period of 26 weeks.
Period: Overall Study
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Started | 175 | 175 | 175 | 178
Full Analysis Set (FAS) | 175 | 175 | 175 | 178
Safety Analysis Set (SAS) | 175 | 175 | 175 | 178
Completed | 169 | 161 | 163 | 170
Not Completed | 6 | 14 | 12 | 8
Not completed — Withdrawal by Subject | 0 | 5 | 5 | 4
Not completed — Lost to Follow-up | 5 | 7 | 5 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Other | 1 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo | Total
Number analyzed (Participants) | 175 | 175 | 175 | 178 | 703
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (11) | 56 (11) | 54 (11) | 54 (11) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 82 | 89 | 89 | 346
  Male | 89 | 93 | 86 | 89 | 357
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race of participants
  Participants
    White | 135 | 131 | 130 | 132 | 528
    Black or African American | 6 | 11 | 10 | 10 | 37
    Asian | 31 | 30 | 29 | 31 | 121
    American Indian or Alaska Native | 1 | 1 | 1 | 1 | 4
    Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 0 | 1
    Other | 2 | 2 | 4 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity of participants
  Participants
    Hispanic or Latino | 52 | 31 | 46 | 51 | 180
    Not Hispanic or Latino | 116 | 133 | 122 | 121 | 492
    Not applicable | 7 | 11 | 7 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) to week 26 in glycosylated haemoglobin (HbA1c). The endpoint was evaluated based on data from the in-trial observation period. The in-trial observation period - time period from when a subject was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product. The primary endpoint was also analysed based on data from the on-treatment without rescue medication observation period. The on-treatment without rescue medication observation period - time period when a subject was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Percentage of HbA1c
  In-trial: number analyzed (Participants) | 167 | 160 | 160 | 168
  In-trial | -0.9 (1.2) | -1.3 (1.0) | -1.5 (1.0) | -0.3 (1.2)
  On-treatment without rescue medication: number analyzed (Participants) | 149 | 146 | 147 | 133
  On-treatment without rescue medication | -0.9 (1.2) | -1.4 (0.9) | -1.6 (1.0) | -0.3 (1.2)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to impute missing data for week 26, assuming that the missing data mechanism was missing at random within the groups used for the imputation. The imputed data sets were analysed using an analysis of covariance (ANCOVA) model with treatment and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any additional anti-diabetic medication for all randomised subjects regardless of premature trial product discontinuation (treatment policy estimand); p < 0.0001, Pattern mixed model — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -1.1, 95% CI 2-sided [-1.3 to -0.9] — Oral Semaglutide 14 mg - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to impute missing data for week 26, assuming that the missing data mechanism was missing at random within the groups used for the imputation. The imputed data sets were analysed using an ANCOVA model with treatment and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixed model — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -0.9, 95% CI 2-sided [-1.1 to -0.6] — Oral Semaglutide 7 mg - Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 3 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixed model — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -0.6, 95% CI 2-sided [-0.8 to -0.4] — Oral Semaglutide 3 mg - Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 3 mg vs Placebo; The analysis was based on a mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment and region as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication (hypothetical estimand); p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -0.7, 95% CI 2-sided [-0.9 to -0.5] — Oral Semaglutide 3 mg - placebo
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -1.2, 95% CI 2-sided [-1.5 to -1.0] — Oral Semaglutide 7 mg - placebo
Statistical Analysis 6: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -1.4, 95% CI 2-sided [-1.7 to -1.2] — Oral Semaglutide 14 mg - placebo

2. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) to week 26 in body weight. The endpoint was evaluated based on data from the in-trial observation period. The in-trial observation period - time period from when a subject was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product. The primary endpoint was also analysed based on data from the on-treatment without rescue medication observation period. The on-treatment without rescue medication observation period - time period when a subject was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
kg
  In-trial: number analyzed (Participants) | 168 | 160 | 160 | 168
  In-trial | -1.5 (3.3) | -2.6 (4.1) | -4.0 (4.2) | -1.4 (3.5)
  On-treatment without rescue medication: number analyzed (Participants) | 150 | 150 | 149 | 134
  On-treatment without rescue medication | -1.8 (3.3) | -2.8 (4.0) | -4.3 (4.2) | -1.6 (3.6)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to impute missing data for week 26, assuming that the missing data mechanism was missing at random within the groups used for the imputation. The imputed data sets were analysed using an ANCOVA model with treatment and region as categorical fixed effects and baseline body weight value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixed model — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -2.3, 95% CI 2-sided [-3.1 to -1.5] — Oral Semaglutide 14 mg - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0866, Pattern mixed model — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -0.9, 95% CI 2-sided [-1.9 to 0.1] — Oral Semaglutide 7 mg - Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 3 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8692, Pattern mixed model — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -0.1, 95% CI 2-sided [-0.9 to 0.8] — Oral Semaglutide 3 mg - Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 3 mg vs Placebo; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment and region as categorical fixed effects and the baseline body weight value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.7075, MMRM; Mean treatment difference = -0.2, 95% CI 2-sided [-1.0 to 0.6] — Oral Semaglutide 3 mg - Placebo
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.0138, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -1.0, 95% CI 2-sided [-1.8 to -0.2] — Oral Semaglutide 7 mg - Placebo
Statistical Analysis 6: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Mean treatment difference = -2.6, 95% CI 2-sided [-3.4 to -1.8] — Oral Semaglutide 14 mg - Placebo

3. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline (week 0) to week 26 in fasting plasma glucose. The endpoint was evaluated based on data from the in-trial observation period. The in-trial observation period - time period from when a subject was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 166 | 160 | 160 | 166
mmol/L | -0.89 (2.67) | -1.52 (2.28) | -1.92 (2.04) | -0.18 (2.37)

4. Secondary Outcome: Change in Mean 7-point SMPG Profile
Description: Change from baseline (week 0) to week 26 in mean 7-point self-measured plasma glucose (SMPG) profile. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 149 | 146 | 141 | 147
mmol/L | -1.8 (2.3) | -2.1 (2.0) | -2.3 (2.4) | -0.5 (2.6)

5. Secondary Outcome: Change in Mean Postprandial Increment Over All Meals in SMPG
Description: Change from baseline (week 0) to week 26 in the average of the post-prandial increments over all meals. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 149 | 148 | 141 | 147
mmol/L | -0.4 (2.3) | -0.8 (2.0) | -1.2 (2.1) | -0.3 (2.0)

6. Secondary Outcome: Change in Fasting Insulin - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in fasting insulin (pmol/L) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting insulin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 157 | 152 | 159 | 163
Ratio of fasting insulin | 1.12 (59.2) | 1.07 (49.2) | 0.98 (45.0) | 0.97 (59.2)

7. Secondary Outcome: Change in Fasting Pro-insulin - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in fasting pro-insulin (pmol/L) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting pro-insulin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 162 | 158 | 156 | 165
Ratio of fasting pro-insulin | 0.84 (71.5) | 0.74 (74.3) | 0.62 (75.5) | 0.89 (76.5)

8. Secondary Outcome: Change in Fasting Glucagon - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in fasting glucagon (pg/mL) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting glucagon
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 161 | 158 | 159 | 163
Ratio of fasting glucagon | 1.00 (28.2) | 0.90 (27.1) | 0.89 (25.7) | 0.95 (25.4)

9. Secondary Outcome: Change in HOMA-IR (Insulin Resistance) - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in homeostatic model assessment index of insulin resistance (HOMA-IR) (%) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-IR
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 156 | 152 | 159 | 161
Ratio of HOMA-IR | 1.00 (74.6) | 0.88 (66.7) | 0.76 (60.4) | 0.92 (75.0)

10. Secondary Outcome: Change in HOMA-B (Beta-cell Function) - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in homeostatic model assessment index of beta-cell function (HOMA-B) (%) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-B
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 156 | 152 | 159 | 160
Ratio of HOMA-B | 1.40 (73.2) | 1.51 (60.5) | 1.60 (58.4) | 1.01 (61.9)

11. Secondary Outcome: Change in CRP - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in C-reactive protein (CRP) (mg/L) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of CRP
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 165 | 159 | 158 | 165
Ratio of CRP | 0.89 (87.5) | 0.72 (118.2) | 0.81 (123.7) | 0.99 (108.3)

12. Secondary Outcome: Change in Body Weight (%)
Description: Change from baseline (week 0) to week 26 in body weight. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 168 | 160 | 160 | 168
Percentage change | -1.67 (4.08) | -2.85 (4.57) | -4.71 (5.00) | -1.37 (3.58)

13. Secondary Outcome: Change in BMI
Description: Change from baseline (week 0) to week 26 in body mass index (BMI). Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 168 | 160 | 160 | 168
kg/m^2 | -0.6 (1.2) | -0.9 (1.5) | -1.5 (1.5) | -0.5 (1.2)

14. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) to week 26 in waist circumference. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 167 | 159 | 158 | 167
cm | -2.0 (4.8) | -2.3 (5.0) | -4.1 (4.9) | -0.9 (4.4)

15. Secondary Outcome: Change in Fasting Total Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in fasting total cholesterol (mmol/L) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting total cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 165 | 159 | 158 | 166
Ratio of fasting total cholesterol | 0.98 (15.6) | 0.98 (18.4) | 0.96 (19.0) | 1.01 (17.9)

16. Secondary Outcome: Change in Fasting LDL Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in fasting low-density lipoprotein (LDL) cholesterol (mmol/L) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting LDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 165 | 159 | 158 | 165
Ratio of fasting LDL cholesterol | 0.95 (27.8) | 0.97 (28.8) | 0.95 (31.6) | 1.00 (26.2)

17. Secondary Outcome: Change in Fasting HDL Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in fasting high-density lipoprotein (HDL) cholesterol (mmol/L) is presented as ratio to baseline. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 165 | 159 | 158 | 166
Ratio of fasting HDL cholesterol | 1.03 (14.6) | 1.05 (14.9) | 1.02 (14.7) | 1.03 (14.0)

18. Secondary Outcome: Change in Fasting Triglycerides - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in triglycerides (mmol/L) is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting triglycerides
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 165 | 159 | 158 | 166
Ratio of fasting triglycerides | 1.01 (35.8) | 0.90 (41.1) | 0.91 (37.8) | 1.00 (39.2)

19. Secondary Outcome: Participants Who Achieve HbA1c < 7.0 % (53 mmol/Mol) ADA Target (Yes/no)
Description: Participants who achieved HbA1c <7.0% (53 mmol/mol) (American Diabetes Association (ADA) target), at week 26 are presented. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 167 | 160 | 160 | 168
Participants
  Yes | 92 | 110 | 123 | 52
  No | 75 | 50 | 37 | 116

20. Secondary Outcome: Participants Who Achieve HbA1c ≤ 6.5 % (48 mmol/Mol) AACE Target (Yes/no)
Description: Participants who achieved HbA1c ≤6.5% (48 mmol/mol) (American Association of Clinical Endocrinologists (AACE) target), at week 26 are presented. The results are based on the data from the in-trial observation period. In trial observation period: the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 167 | 160 | 160 | 168
Participants
  Yes | 60 | 76 | 102 | 30
  No | 107 | 84 | 58 | 138

21. Secondary Outcome: Participants Who Achieve Body Weight Loss ≥ 5 % (Yes/no)
Description: Participants who achieved body weight loss more than or equal to 5% of their baseline body weight (yes/no) at week 26 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 168 | 160 | 160 | 168
Participants
  Yes | 33 | 43 | 66 | 25
  No | 135 | 117 | 94 | 143

22. Secondary Outcome: Participants Who Achieve Body Weight Loss ≥ 10 % (Yes/no)
Description: Participants who achieved body weight loss more than or equal to 10% of their baseline body weight (yes/no) at week 26 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 168 | 160 | 160 | 168
Participants
  Yes | 4 | 13 | 23 | 2
  No | 164 | 147 | 137 | 166

23. Secondary Outcome: Participants Who Achieve HbA1c < 7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG-confirmed Symptomatic Hypoglycaemia) and Without Body Weight Gain (Yes/no)
Description: Participants who achieved HbA1c less than 7.0 % without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) at week 26 are presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 167 | 160 | 160 | 168
Participants
  Yes | 62 | 91 | 110 | 39
  No | 105 | 69 | 50 | 129

24. Secondary Outcome: Participants Who Achieve HbA1c Reduction ≥ 1.0% (10.9 mmol/Mol) and Weight Loss ≥ 3% (Yes/no)
Description: Participants who achieved HbA1c reduction more than or equal to 1% of their baseline HbA1c and weight loss of more than or equal to 3% of their baseline body weight (yes/no) at week 26 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 167 | 160 | 160 | 168
Participants
  Yes | 30 | 59 | 81 | 18
  No | 137 | 101 | 79 | 150

25. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the period from week 0 to week 26. Additional anti-diabetic medication was defined as any new anti-diabetic medication used for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment (week 26), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Participants | 16 | 8 | 7 | 35
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment and region as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0043, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.26 to 0.78] — Oral Semaglutide 3 mg / Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 25, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0002, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.18 to 0.59] — Oral Semaglutide 7 mg / Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 25, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0002, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.19 to 0.60] — Oral Semaglutide 14 mg / Placebo

26. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the period from week 0 to week 26. Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 0) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication or premature trial product discontinuation.
Time Frame: Weeks 0-26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Participants | 13 | 4 | 2 | 27
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0300, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.25 to 0.93] — Oral Semaglutide 3 mg / Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 26, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.04 to 0.36] — Oral Semaglutide 7 mg / Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 26, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.06, 95% CI 2-sided [0.01 to 0.26] — Oral Semaglutide 14 mg /Placebo

27. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 31 (26-week treatment period + 5-week follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Approximately upto week 31
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Events | 290 | 258 | 304 | 263

28. Secondary Outcome: Change in Amylase - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in amylase (units/litre (U/L)) is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 159 | 152 | 149 | 154
Ratio | 1.05 (21.1) | 1.09 (21.4) | 1.12 (20.2) | 0.99 (25.5)

29. Secondary Outcome: Change in Lipase - Ratio to Baseline
Description: Change from baseline (week 0) to week 26 in lipase (U/L) is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 159 | 152 | 149 | 154
Ratio | 1.14 (43.8) | 1.27 (51.1) | 1.33 (45.1) | 0.99 (54.2)

30. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at week 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 161 | 154 | 151 | 158
beats/min | 0 (9) | 1 (9) | 3 (9) | 1 (9)

31. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change from baseline (week 0) in SBP was evaluated at week 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 161 | 154 | 151 | 158
mmHg | -3 (14) | -5 (13) | -5 (14) | -3 (14)

32. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: Change from baseline (week 0) in DBP was evaluated at week 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 161 | 154 | 151 | 158
mmHg | -1 (9) | -2 (8) | -1 (9) | -1 (9)

33. Secondary Outcome: Change in Electrocardiogram (ECG) Evaluation
Description: Change from baseline (week 0) in ECG was evaluated at week 26. Change from baseline results are presented as shift in findings (normal, abnormal and not clinically significant (NCS) and abnormal and clinically significant (CS)) from week 0 to week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 114 | 102 | 100 | 110
  Normal (week 0) to normal (week 26) | 102 | 88 | 96 | 97
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 114 | 102 | 100 | 110
  Normal (week 0) to abnormal NCS (week 26) | 11 | 13 | 4 | 13
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 114 | 102 | 100 | 110
  Normal (week 0) to abnormal CS (week 26) | 1 | 1 | 0 | 0
  Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 52 | 52 | 59 | 54
  Abnormal NCS (week 0) to normal (week 26) | 12 | 12 | 20 | 14
  Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 52 | 52 | 59 | 54
  Abnormal NCS (week 0) to abnormal NCS (week 26) | 40 | 39 | 39 | 40
  Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 52 | 52 | 59 | 54
  Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 1 | 0 | 0
  Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 1 | 5 | 0 | 2
  Abnormal CS (week 0) to normal (week 26) | 0 | 1 | 0 | 0
  Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 1 | 5 | 0 | 2
  Abnormal CS (week 0) to abnormal NCS (week 26) | 1 | 3 | 0 | 2
  Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 1 | 5 | 0 | 2
  Abnormal CS (week 0) to abnormal CS (week 26) | 0 | 1 | 0 | 0

34. Secondary Outcome: Change in Physical Examination
Description: Participants with physical examination findings, normal, abnormal NCS and abnormal CS at baseline (week -2) and week 26 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product. Results are presented for the following examinations: 1) Cardiovascular system; 2) Nervous system (central and peripheral); 3) Gastrointestinal system, incl. mouth; 4) General appearance; 5) Head (ears, eyes, nose), throat, neck; 6) Lymph node palpation; 7) Musculoskeletal system; 8) Respiratory system; 9) Skin; 10) Thyroid gland.
Time Frame: Week 0, week 26
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Participants
  1) Cardiovascular system (week -2): Normal | 163 | 167 | 167 | 172
  1) Cardiovascular system (week -2): Abnormal NCS | 12 | 8 | 8 | 6
  1) Cardiovascular system (week -2): Abnormal CS | 0 | 0 | 0 | 0
  1) Cardiovascular system (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  1) Cardiovascular system (week 26): Normal | 157 | 149 | 155 | 162
  1) Cardiovascular system (week 26): Abnormal NCS | 10 | 9 | 4 | 4
  1) Cardiovascular system (week 26): Abnormal CS | 0 | 1 | 0 | 1
  2) Central and peripheral nervous system (week -2): Normal | 165 | 171 | 168 | 169
  2) Central and peripheral nervous system (week -2): Abnormal NCS | 10 | 4 | 7 | 9
  2) Central and peripheral nervous system (week -2): Abnormal CS | 0 | 0 | 0 | 0
  2) Central and peripheral nervous system (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  2) Central and peripheral nervous system (week 26): Normal | 157 | 157 | 153 | 159
  2) Central and peripheral nervous system (week 26): Abnormal NCS | 10 | 2 | 6 | 8
  2) Central and peripheral nervous system (week 26): Abnormal CS | 0 | 0 | 0 | 0
  3) Gastrointestinal system, incl. mouth (week -2): Normal | 164 | 169 | 159 | 168
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal NCS | 11 | 6 | 16 | 10
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal CS | 0 | 0 | 0 | 0
  3) Gastrointestinal system, incl. mouth (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  3) Gastrointestinal system, incl. mouth (week 26): Normal | 153 | 154 | 148 | 157
  3) Gastrointestinal system, incl. mouth (week 26): Abnormal NCS | 13 | 5 | 11 | 10
  3) Gastrointestinal system, incl. mouth (week 26): Abnormal CS | 1 | 0 | 0 | 0
  4) General appearance (week -2): Normal | 143 | 152 | 153 | 157
  4) General appearance (week -2): Abnormal NCS | 32 | 23 | 20 | 21
  4) General appearance (week -2): Abnormal CS | 0 | 0 | 2 | 0
  4) General appearance (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  4) General appearance (week 26): Normal | 138 | 141 | 141 | 148
  4) General appearance (week 26): Abnormal NCS | 29 | 17 | 17 | 19
  4) General appearance (week 26): Abnormal CS | 0 | 1 | 1 | 0
  5) Head, ears, eyes, nose, throat, neck (week -2): Normal | 163 | 165 | 165 | 168
  5) Head, ears, eyes, nose, throat, neck (week -2): Abnormal NCS | 12 | 10 | 10 | 9
  5) Head, ears, eyes, nose, throat, neck (week -2): Abnormal CS | 0 | 0 | 0 | 1
  5) Head, ears, eyes, nose, throat, neck (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  5) Head, ears, eyes, nose, throat, neck (week 26): Normal | 155 | 149 | 149 | 155
  5) Head, ears, eyes, nose, throat, neck (week 26): Abnormal NCS | 12 | 10 | 10 | 11
  5) Head, ears, eyes, nose, throat, neck (week 26): Abnormal CS | 0 | 0 | 0 | 1
  6) Lymph node palpation (week -2): Normal | 175 | 175 | 175 | 178
  6) Lymph node palpation (week -2): Abnormal NCS | 0 | 0 | 0 | 0
  6) Lymph node palpation (week -2): Abnormal CS | 0 | 0 | 0 | 0
  6) Lymph node palpation (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  6) Lymph node palpation (week 26): Normal | 167 | 159 | 159 | 167
  6) Lymph node palpation (week 26): Abnormal NCS | 0 | 0 | 0 | 0
  6) Lymph node palpation (week 26): Abnormal CS | 0 | 0 | 0 | 0
  7) Musculoskeletal system (week -2): Normal | 164 | 169 | 167 | 167
  7) Musculoskeletal system (week -2): Abnormal NCS | 11 | 6 | 8 | 11
  7) Musculoskeletal system (week -2): Abnormal CS | 0 | 0 | 0 | 0
  7) Musculoskeletal system (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  7) Musculoskeletal system (week 26): Normal | 155 | 154 | 152 | 157
  7) Musculoskeletal system (week 26): Abnormal NCS | 11 | 5 | 6 | 10
  7) Musculoskeletal system (week 26): Abnormal CS | 1 | 0 | 1 | 0
  8) Respiratory system (week -2): Normal | 173 | 172 | 173 | 174
  8) Respiratory system (week -2): Abnormal NCS | 2 | 3 | 2 | 4
  8) Respiratory system (week -2): Abnormal CS | 0 | 0 | 0 | 0
  8) Respiratory system (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  8) Respiratory system (week 26): Normal | 163 | 157 | 159 | 166
  8) Respiratory system (week 26): Abnormal NCS | 4 | 2 | 0 | 1
  8) Respiratory system (week 26): Abnormal CS | 0 | 0 | 0 | 0
  9) Skin (week -2): Normal | 137 | 156 | 150 | 150
  9) Skin (week -2): Abnormal NCS | 36 | 18 | 24 | 27
  9) Skin (week -2): Abnormal CS | 2 | 1 | 1 | 1
  9) Skin (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  9) Skin (week 26): Normal | 136 | 145 | 140 | 140
  9) Skin (week 26): Abnormal NCS | 30 | 13 | 18 | 24
  9) Skin (week 26): Abnormal CS | 1 | 1 | 1 | 3
  10) Thyroid gland (week -2): Normal | 173 | 170 | 169 | 176
  10) Thyroid gland (week -2): Abnormal NCS | 1 | 4 | 6 | 2
  10) Thyroid gland (week -2): Abnormal CS | 1 | 1 | 0 | 0
  10) Thyroid gland (week 26): number analyzed (Participants) | 167 | 159 | 159 | 167
  10) Thyroid gland (week 26): Normal | 165 | 155 | 156 | 165
  10) Thyroid gland (week 26): Abnormal NCS | 1 | 4 | 3 | 2
  10) Thyroid gland (week 26): Abnormal CS | 1 | 0 | 0 | 0

35. Secondary Outcome: Change in Eye Examination Category
Description: Participants with eye examination (fundoscopy) findings, normal, abnormal NCS and abnormal CS at baseline (week -2), and week 26 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Participants
  Left eye (week -2): number analyzed (Participants) | 173 | 175 | 175 | 178
  Left eye (week -2): Normal | 109 | 112 | 109 | 122
  Left eye (week -2): Abnormal NCS | 59 | 59 | 63 | 54
  Left eye (week -2): Abnormal CS | 5 | 4 | 3 | 2
  Left eye (week 26): number analyzed (Participants) | 158 | 153 | 156 | 162
  Left eye (week 26): Normal | 101 | 94 | 99 | 105
  Left eye (week 26): Abnormal NCS | 55 | 55 | 54 | 54
  Left eye (week 26): Abnormal CS | 2 | 4 | 3 | 3
  Right eye (week -2): number analyzed (Participants) | 174 | 175 | 175 | 178
  Right eye (week -2): Normal | 111 | 116 | 108 | 120
  Right eye (week -2): Abnormal NCS | 58 | 55 | 63 | 55
  Right eye (week -2): Abnormal CS | 5 | 4 | 4 | 3
  Right eye (week 26): number analyzed (Participants) | 157 | 153 | 156 | 162
  Right eye (week 26): Normal | 103 | 93 | 98 | 106
  Right eye (week 26): Abnormal NCS | 52 | 56 | 55 | 53
  Right eye (week 26): Abnormal CS | 2 | 4 | 3 | 3

36. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide binding antibodies anytime during post-baseline visits (week 0 to week 31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 173 | 171 | 172
Participants | 2 | 1 | 0

37. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide neutralising antibodies anytime during post-baseline visits (week 0 to week 31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 173 | 171 | 172
Participants | 1 | 0 | 0

38. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide binding antibodies cross reacting with native glucagon-like peptide-1 (GLP-1) anytime during post-baseline visits (week 0 to week 31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 173 | 171 | 172
Participants | 2 | 1 | 0

39. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Number of participants who measured with anti-semaglutide neutralising antibodies cross reacting with native GLP-1 anytime during post-baseline visits (week 0 to week 31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 173 | 171 | 172
Participants | 0 | 0 | 0

40. Secondary Outcome: Anti-semaglutide Binding Antibody Levels
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). It is based on the data from participants who were measured with anti-semaglutide antibodies anytime during post-baseline visits (week 0 to week 31). Results are presented as percentage of bound radioactivity-labelled semaglutide /total added radioactivity-labelled semaglutide (%B/T). Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analysed = participants who were found positive for anti-semaglutide antibodies.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 2 | 1 | 0
%B/T
  Week 4 | 15 (13) | 2 (0) |
  Week 8: number analyzed (Participants) | 2 | 0 | 0
  Week 8 | 7 (4) |  |
  Week 14: number analyzed (Participants) | 0 | 1 | 0
  Week 14 |  | 3 (0) |
  Week 26: number analyzed (Participants) | 0 | 0 | 0
  Week 31: number analyzed (Participants) | 1 | 0 | 0
  Week 31 | 3 (0) |  |

41. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes During Exposure to Trial Product
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during week 0 to week 31 (26-weeks treatment period + 5-weeks follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Episodes | 5 | 2 | 1 | 1

42. Secondary Outcome: Participants With Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes During Exposure to Trial Product
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded from week 0 to week 31 (26-week treatment period + 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-31
Population: as for outcome 41
Measure: Number; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Participants | 5 | 2 | 1 | 1

43. Secondary Outcome: SNAC Plasma Concentrations
Description: This outcome measure is only applicable for the oral semaglutide 3 mg, 7 mg and 14 mg treatment arms. Sodium N-[8-(2-hydroxybenzoyl) amino]caprylate (SNAC) plasma concentrations were measured after 25 and 40 minutes post-dose at weeks 4, 14 and 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 175 | 175 | 175
Nanograms per milliliter (ng/mL)
  Week 4: 25 minutes post-dose: number analyzed (Participants) | 169 | 166 | 168
  Week 4: 25 minutes post-dose | 443.5 (378.4) | 446.0 (329.4) | 449.4 (330.5)
  Week 4: 40 minutes post-dose: number analyzed (Participants) | 169 | 167 | 168
  Week 4: 40 minutes post-dose | 381.7 (227.5) | 367.3 (238.5) | 387.7 (186.3)
  Week 14: 25 minutes post-dose: number analyzed (Participants) | 165 | 158 | 153
  Week 14: 25 minutes post-dose | 384.6 (415.4) | 380.6 (427.0) | 338.2 (339.5)
  Week 14: 40 minutes post-dose: number analyzed (Participants) | 165 | 155 | 154
  Week 14: 40 minutes post-dose | 361.0 (259.2) | 326.4 (350.1) | 262.2 (377.4)
  Week 26: 25 minutes post-dose: number analyzed (Participants) | 159 | 152 | 149
  Week 26: 25 minutes post-dose | 412.4 (533.3) | 479.6 (334.3) | 330.9 (578.4)
  Week 26: 40 minutes post-dose: number analyzed (Participants) | 159 | 151 | 148
  Week 26: 40 minutes post-dose | 299.1 (411.1) | 401.0 (271.6) | 300.9 (372.5)

44. Secondary Outcome: Semaglutide Plasma Concentrations for Population PK Analysis
Description: This outcome measure is only applicable for the oral semaglutide 3 mg, 7 mg and 14 mg treatment arms. Semaglutide plasma concentrations were measured at weeks 4, 8, 14 and 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0 - 26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per litre (nmol/L)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 175 | 175 | 175
Nanomoles per litre (nmol/L)
  Week 4: number analyzed (Participants) | 168 | 169 | 169
  Week 4 | 3.120 (130.2) | 2.765 (118.7) | 2.829 (127.6)
  Week 8: number analyzed (Participants) | 170 | 162 | 161
  Week 8 | 3.073 (132.0) | 6.216 (158.5) | 6.461 (164.3)
  Week 14: number analyzed (Participants) | 163 | 158 | 154
  Week 14 | 2.716 (145.7) | 6.375 (177.3) | 12.69 (235.2)
  Week 26: number analyzed (Participants) | 160 | 151 | 151
  Week 26 | 2.466 (158.7) | 5.016 (195.3) | 11.07 (252.6)

45. Secondary Outcome: Change in SF-36v2 (Acute Version) Health Survey: Scores From the 8 Domains, the Physical Component Summary (PCS) and the Mental Component Summary (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the sub-domain scores and component summary (PCS and MCS) scores were evaluated at week 26. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 165 | 158 | 158 | 167
Score on a scale
  1) Physical Functioning | 0.14 (6.25) | 1.18 (6.36) | 1.05 (5.75) | 0.66 (6.18)
  2) Role-Physical | -0.41 (6.62) | -0.08 (7.04) | 0.79 (6.86) | -0.25 (6.73)
  3) Bodily Pain | 1.17 (9.02) | -0.67 (9.37) | -0.14 (9.61) | 0.40 (8.77)
  4) General Health | 0.97 (8.08) | 0.92 (7.51) | 2.07 (6.88) | 0.18 (7.53)
  5) Vitality | -0.08 (8.10) | 0.77 (7.83) | 0.40 (8.21) | -0.47 (8.02)
  6) Social Functioning | 0.21 (9.15) | 1.00 (7.64) | 0.88 (7.94) | 0.18 (8.37)
  7) Role-Emotional | -0.05 (9.89) | -0.63 (9.27) | 0.85 (9.49) | -1.28 (10.02)
  8) Mental Health | 0.04 (7.62) | 0.06 (8.51) | 0.67 (8.74) | -0.25 (9.64)
  Physical component summary | 0.52 (6.04) | 0.61 (5.86) | 0.89 (5.66) | 0.65 (5.44)
  Mental component summary | -0.07 (8.08) | -0.00 (8.00) | 0.67 (8.40) | -0.90 (9.08)

46. Secondary Outcome: IWQOL-Lite Clinical Trial Version: Total Score of the 22 Items (Used for Validation of the Questionnaire)
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on patients' quality of life within the context of clinical trials. IWQOL-Lite-CT is a 22-item questionnaire-based instrument used to assess the impact of body weight changes on participant's overall health-related quality of life (HRQoL). All IWQOL-Lite-CT composite scores range from 0 to 100, with higher scores reflecting better levels of functioning. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Score on a scale
  1) Trouble bending over: number analyzed (Participants) | 165 | 158 | 158 | 167
  1) Trouble bending over | -0.17 (1.09) | -0.12 (1.07) | -0.13 (0.96) | -0.08 (1.06)
  2) Tired/winded walking up stairs: number analyzed (Participants) | 165 | 158 | 158 | 167
  2) Tired/winded walking up stairs | -0.13 (1.03) | -0.16 (1.04) | -0.23 (1.02) | -0.11 (0.96)
  3) Difficulty standing: number analyzed (Participants) | 164 | 158 | 157 | 167
  3) Difficulty standing | -0.12 (1.34) | -0.22 (1.40) | -0.08 (1.18) | -0.01 (1.28)
  4) Uncomfortable in small seats: number analyzed (Participants) | 164 | 158 | 158 | 165
  4) Uncomfortable in small seats | -0.09 (1.08) | -0.05 (1.20) | -0.09 (1.04) | 0.03 (1.33)
  5) Bodily pain: number analyzed (Participants) | 165 | 158 | 158 | 167
  5) Bodily pain | -0.27 (1.10) | -0.08 (1.11) | -0.06 (1.05) | -0.14 (1.07)
  6) Self-conscious eating in social settings: number analyzed (Participants) | 165 | 157 | 158 | 166
  6) Self-conscious eating in social settings | 0.00 (0.97) | 0.01 (1.15) | -0.11 (0.96) | -0.10 (1.08)
  7) Less confident: number analyzed (Participants) | 164 | 157 | 158 | 167
  7) Less confident | -0.22 (1.05) | -0.29 (0.98) | -0.35 (1.00) | -0.20 (1.07)
  8) Feel judged by others: number analyzed (Participants) | 165 | 158 | 158 | 167
  8) Feel judged by others | -0.01 (1.00) | -0.23 (0.92) | -0.20 (0.93) | -0.13 (0.90)
  9) Less important/worthy of respect: number analyzed (Participants) | 165 | 158 | 158 | 167
  9) Less important/worthy of respect | -0.05 (0.83) | -0.04 (0.79) | -0.11 (0.74) | -0.15 (0.77)
  10) Frustrated shopping for clothes: number analyzed (Participants) | 165 | 158 | 155 | 167
  10) Frustrated shopping for clothes | -0.08 (0.95) | -0.10 (0.96) | -0.19 (0.92) | -0.14 (1.09)
  11) Feel bad or upset in pictures: number analyzed (Participants) | 165 | 158 | 158 | 167
  11) Feel bad or upset in pictures | -0.16 (1.07) | -0.20 (0.91) | -0.23 (0.99) | -0.14 (1.07)
  12) Feel down or depressed: number analyzed (Participants) | 165 | 157 | 158 | 167
  12) Feel down or depressed | -0.22 (1.07) | -0.18 (0.88) | -0.24 (0.86) | -0.16 (1.01)
  13) Less interested in sex: number analyzed (Participants) | 164 | 157 | 158 | 166
  13) Less interested in sex | -0.14 (1.24) | 0.04 (1.07) | -0.03 (1.11) | -0.06 (1.16)
  14) Avoid social gatherings: number analyzed (Participants) | 164 | 158 | 157 | 167
  14) Avoid social gatherings | 0.05 (0.76) | -0.07 (0.69) | -0.04 (0.63) | -0.02 (0.58)
  15) Less productive: number analyzed (Participants) | 165 | 158 | 158 | 167
  15) Less productive | -0.09 (1.00) | -0.13 (0.97) | -0.10 (0.97) | -0.07 (0.80)
  16) Lack energy to do things I would like to do: number analyzed (Participants) | 165 | 157 | 156 | 167
  16) Lack energy to do things I would like to do | -0.14 (1.06) | -0.20 (1.11) | -0.14 (1.01) | -0.03 (1.01)
  17) Not as physically active: number analyzed (Participants) | 165 | 158 | 157 | 167
  17) Not as physically active | -0.09 (1.06) | -0.41 (1.26) | -0.04 (1.11) | -0.08 (1.22)
  18) Unable to walk far/quickly: number analyzed (Participants) | 165 | 158 | 158 | 167
  18) Unable to walk far/quickly | -0.08 (1.09) | -0.29 (1.26) | 0.02 (0.99) | -0.19 (1.21)
  19) Worried about health: number analyzed (Participants) | 165 | 157 | 158 | 167
  19) Worried about health | -0.32 (1.35) | -0.49 (1.39) | -0.42 (1.27) | -0.30 (1.39)
  20) Limited self-esteem: number analyzed (Participants) | 164 | 158 | 158 | 166
  20) Limited self-esteem | -0.03 (1.04) | -0.09 (1.10) | -0.07 (1.02) | -0.09 (0.89)
  21) Self-conscious about weight: number analyzed (Participants) | 165 | 158 | 158 | 167
  21) Self-conscious about weight | -0.10 (0.92) | -0.12 (1.06) | 0.01 (1.08) | -0.05 (0.91)
  22) Frustrated/upset with self: number analyzed (Participants) | 165 | 157 | 157 | 167
  22) Frustrated/upset with self | -0.12 (0.91) | -0.25 (1.02) | -0.14 (1.08) | 0.02 (0.91)

47. Secondary Outcome: PGI-S Item: Scores of the Two Individual Items (Used for Validation of the IWQOL Questionnaire)
Description: Patient global impression of status (PGI-S) is a 2-item questionnaire used to assess the participant's impression of physical functioning and mental health status during the clinical trial. The PGI-S contains two items evaluated on a 5-point graded response scale. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 175 | 175 | 175 | 178
Participants
  1) Physical functioning status: number analyzed (Participants) | 167 | 157 | 159 | 167
  1) Physical functioning status: Poor | 6 | 11 | 11 | 7
  1) Physical functioning status: Fair | 50 | 51 | 45 | 59
  1) Physical functioning status: Good | 67 | 53 | 56 | 71
  1) Physical functioning status: Very good | 30 | 38 | 32 | 23
  1) Physical functioning status: Excellent | 14 | 4 | 15 | 7
  2) Emotional status: number analyzed (Participants) | 167 | 158 | 159 | 166
  2) Emotional status: Poor | 10 | 7 | 9 | 9
  2) Emotional status: Fair | 41 | 41 | 38 | 42
  2) Emotional status: Good | 62 | 51 | 55 | 59
  2) Emotional status: Very good | 32 | 48 | 33 | 41
  2) Emotional status: Excellent | 22 | 11 | 24 | 15

48. Secondary Outcome: PGI-C Item: Scores of the Two Individual Items (Used for Validation of the IWQOL Questionnaire)
Description: Patient global impression of change (PGI-C) is a 2-item questionnaire used to assess the participant's impression of change from baseline in physical functioning and mental health status. The PGI-C contains two items evaluated on a 7-point graded response scale. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 167 | 158 | 159 | 167
Participants
  1) Physical functioning change: Much worse | 0 | 0 | 1 | 1
  1) Physical functioning change: Moderately worse | 1 | 2 | 0 | 1
  1) Physical functioning change: A little worse | 6 | 2 | 3 | 3
  1) Physical functioning change: No difference | 56 | 44 | 29 | 66
  1) Physical functioning change: A little better | 45 | 42 | 48 | 36
  1) Physical functioning change: Moderately better | 23 | 28 | 31 | 31
  1) Physical functioning change: Much better | 36 | 40 | 47 | 29
  2) Emotional change: Much worse | 1 | 0 | 1 | 0
  2) Emotional change: Moderately worse | 0 | 0 | 0 | 1
  2) Emotional change: A little worse | 5 | 2 | 3 | 2
  2) Emotional change: No difference | 60 | 53 | 36 | 63
  2) Emotional change: A little better | 38 | 32 | 37 | 39
  2) Emotional change: Moderately better | 18 | 27 | 32 | 32
  2) Emotional change: Much better | 45 | 44 | 50 | 30

ADVERSE EVENTS:
Time Frame: Week 0 to week 31 (26 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/175 | 1/175 | 0/178
Serious Adverse Events (participants affected / at risk) | 5/175 | 3/175 | 2/175 | 8/178
Other Adverse Events (participants affected / at risk) | 48/175 | 37/175 | 45/175 | 26/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=175) | Oral Semaglutide 7 mg (N=175) | Oral Semaglutide 14 mg (N=175) | Placebo (N=178)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcitonin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palatoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=175) | Oral Semaglutide 7 mg (N=175) | Oral Semaglutide 14 mg (N=175) | Placebo (N=178)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 9 (9) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (18) | 9 (9) | 9 (10) | 4 (4)
Headache (Nervous system disorders) | 6 (7) | 10 (16) | 9 (31) | 9 (12)
Influenza (Infections and infestations) | 9 (9) | 5 (5) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (11) | 11 (11) | 3 (4) | 6 (7)
Nausea (Gastrointestinal disorders) | 14 (17) | 9 (13) | 28 (43) | 10 (12)
Vomiting (Gastrointestinal disorders) | 5 (5) | 8 (11) | 12 (15) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT02906930/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT02906930/SAP_001.pdf